CLINICAL TRIAL: NCT05456048
Title: Influence of Molecular Abnormalities on Treatment Response of the Regimen of Venetoclax Plus Azacytidine Combined With Homoharringtonine Versus Venetoclax Plus Hypomethylating Agents (HMA) in Relapsed/Refractory Acute Myeloid Leukemia
Brief Title: Influence of Molecular Abnormalities on Response of VAH vs. VEN+HMA in RR-AML
Status: Completed | Type: Observational
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Collaborators: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other); Zhongshan People's Hospital, Guangdong, China (Other); Shenzhen Hospital of Southern Medical University (Other); Peking University Shenzhen Hospital (Other); Shenzhen Second People's Hospital (Other); The Seventh Affiliated Hospital of Sun Yat-sen University (Other); Southern Medical University, China (Other); First People's Hospital of Chenzhou (Other); First Affiliated Hospital of Guangxi Medical University (Other)
Responsible Party: Principal Investigator, Qifa Liu, Professor, Nanfang Hospital, Southern Medical University
Other Study IDs: VAH-AML-2022
Record Dates: First submitted 2022-07-03; First posted 2022-07-13 (Actual); Last update posted 2022-07-13 (Actual); Status verified 2022-07

CONDITIONS: Relapsed Acute Myeloid Leukemia; Refractory Acute Myeloid Leukemia; Gene Abnormality; Cytogenetic Abnormality
Keywords: Acute myeloid leukemia; Relapsed/refractory; Gene mutation; Venetoclax; Homoharringtonine
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Chromosome Aberrations; Recurrence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Bone marrow and/or peripheral blood were taken from participants upon enrollment for diagnosis and detection of gene mutations and co-mutations via PCR, direct sequencing and /or next generation sequencing.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- VAH group: Patients assigned to this group received one to two cycles of VAH regimen as salvage therapy of RR-AML.
  Interventions: Drug: VAH regimen
- VEN+HMA group: Patients assigned to this group received one to two cycles of venetoclax plus HMA regimen as salvage therapy of RR-AML.
  Interventions: Drug: VEN+HMA regimen

INTERVENTIONS:
Drug: VAH regimen — VEN was prescribed as 100mg day 1, 200mg day 2, 400mg day 3-14; AZA was used at the dose of 75 mg/m2, day 1-7; HHT was given at a dose of 1mg/m2, day 1-7. The dose of VEN was reduced to 100mg/d if co-administered with posaconazole or voriconazole.
  Groups: VAH group
Drug: VEN+HMA regimen — VEN was prescribed as 100mg day 1, 200mg day 2, 400mg day 3-28; AZA was used at the dose of 75 mg/m2, day 1-7 or DEC 20mg/m2 day 1-5. The dose of VEN was reduced to 100mg/d if co-administered with posaconazole or voriconazole.
  Groups: VEN+HMA group

SUMMARY:
The aim of this study is to reveal the influence of gene mutations on the treatment response of the regimen of HHT combined with Venetoclax plus AZA versus venetoclax plus HMA in the salvage therapy of RR-AML.

DETAILED DESCRIPTION:
Venetoclax-based regimens have heen used in the salvage therapy of relapsed/resfractory (RR) acute myeloid leukemia (AML). More and more studies have shown that molecular abnormalities and venetoclax combined regimens significantly impact the response of venetoclax-based therapy. Our exploratory study revealed that venetoclax plus azacytidine combined with homoharringtonine (VAH) had remarkably higher response than venetoclax plus hypomethylating agents (HMA) in RR-AML. Yet the influence of molecular abnormalities on the response of VAH regimen remains unknown.

ELIGIBILITY:
Inclusion Criteria:

1. RR-AML
2. Patients must have been treated for at least one cycle of VEN-based regimen and finished outcome assessment.

Exclusion Criteria:

1. Acute promyelocytic leukemia (AML subtype M3)
2. Previous exposure to the treatment of VEN-based regimen
3. Cardiac dysfunction (particularly congestive heart failure, unstable coronary artery disease and serious cardiac ventricular arrhythmias requiring antiarrhythmic therapy)
4. Respiratory failure (PaO2 ≤60mmHg)
5. Hepatic abnormalities (total bilirubin ≥2 times the upper limit of normal [ULN], alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≥2 times the ULN)
6. Renal dysfunction (creatinine ≥2 times the ULN or creatinine clearance rate < 30 mL/min)
7. ECOG performance status 3, 4 or 5
8. Substantial history of neurological, psychiatric, endocrine, metabolic, immunological, or any other medical condition not suitable for the trial (investigators' decision)
9. Active acute or chronic graft-versus-host disease (GVHD). Active acute GVHD or chronic GVHD is defined as GVHD requiring either at least 1 mg/kg per day of prednisone (or equivalent) or treatment beyond systemic corticosteroids.
10. Patients with pregnancy
11. Uncontrolled active infection
12. Clinically significant coagulation abnormalities

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cases included in this study were from 3 previous studies of our study group, including 1 exploratory and 2 prospective studies.
Sampling Method: Non-Probability Sample
Enrollment: 231 (Actual)
Dates: Start 2018-12-03 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
CR/CRi | At the end of Cycle 2 (each cycle is 28 days)
  Complete remission and CR with incomplete count recovery

SECONDARY OUTCOMES:
MRD negative | At the end of Cycle 2 (each cycle is 28 days)
  MRD was detected with FCM and defined negative as a ratio < 0.1%
Overall response | At the end of Cycle 2 (each cycle is 28 days)
  Overall response included CR/CRi, MLFS and PR.
Overall survival | 2 years
  The time from enrolling to death or the last follow up
Event-free survival | 2 years
  The time from enrolling to no response, relapse, death or the last follow up

CONTACTS AND LOCATIONS:
Overall Officials: Liu Qifa, MD, Principal Investigator — Nanfang Hospital, Southern Medical University
Locations (1):
- Department of Hematology,Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong, China